CLINICAL TRIAL: NCT00356655
Title: A COHORT AND INTERVENTION STUDY EVALUATING ANTIDEPRESSANT EPIDEMIOLOGY AND ADHERENCE: The ACHIEVA Study
Brief Title: The ACHIEVA Study of Enhanced Pharmacist Care on Antidepressant Use and Response
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: University of Alberta (Other)
Collaborators: Institute of Health Economics, Canada (Other); Dalhousie University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-Gardner
Record Dates: First submitted 2006-07-24; First posted 2006-07-26 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2008-05

CONDITIONS: Depressive Disorder
Keywords: Depressive disorder; Patient compliance; Antidepressive Agents; Patient education; Community pharmacy services; Counseling
MeSH Terms: conditions — Depressive Disorder; Patient Compliance

INTERVENTIONS:
Behavioral: Psychoeducation

SUMMARY:
This a comparative study of enhanced pharmacist care and regular care of patients starting on antidepressants. When providing participants with enhanced care pharmacists will use the Health Professional's Antidepressant Communications Tool (Health PACT) a minimum of three times during face-to-face discussions. This tool was developed specifically for this study. All participants will be followed for 26 weeks and will be assessed for duration of use of their antidepressant, adherence to treatment, and clinical response.

DETAILED DESCRIPTION:
This proposal describes a combined observational study (Phase I) and randomized controlled trial (Phase II). The primary aim of the observational study is to determine the disorders, in particular the types of depression, for which family physicians prescribe antidepressants. The primary aim of the randomized controlled trial (RCT) is to compare the effect of a brief psycho-educational intervention by pharmacists with usual care on antidepressant persistence.

Subjects (n=621 phase 1, n=106 phase 2) will be patients presenting to a pharmacy in Edmonton with a prescription for an antidepressant from a family physician and meeting the following criteria: no antidepressants taken in the preceding six months; 18 years of age or older, and fluent in English. Subjects will be interviewed using modified versions of the depression, generalized anxiety disorder and panic disorder sections of the Diagnostic Interview Schedule; the Beck Depression Inventory; the Beck Anxiety Inventory; and a question on recent stressful life events. For Phase 1 the proportion of subjects with the following DSM-IV diagnoses will be estimated: major depression, "minor depression," generalized anxiety disorder, panic disorder; minor depression will be categorized into "adjustment disorder with depressed mood" and "adjustment disorder with mixed anxiety and depressed mood". The family doctor will be contacted and asked for the diagnosis that prompted the antidepressant prescription.

Subjects with DSM IV depression will be invited to participate in Phase 2. Individuals will be randomized to a pharmacist intervention with the Health PACT, or to usual care. Using the newly-developed Antidepressant Compliance Questionnaire, information on predictors of adherence will be collected at the baseline interview. At weeks 4, 8, 16 and 26, subjects will be contacted by phone and questioned on antidepressant adherence and persistence. At week 8 (or the exit interview if a subject leaves the study early), we will administer the Beck Depression Inventory and the Beck Anxiety Inventory. The primary outcome is treatment persistence, defined as the time to stop antidepressant use. Adherence, defined by the medication possession ratio (MPR), will be also be measured.

ELIGIBILITY:
Inclusion Criteria:

* patient presents to a pharmacy with a prescription for an antidepressant from a family physician
* patient with DSM-IV major or minor depression
* patient has not taken an antidepressant in the preceding six months
* patient is 18 years of age or older
* patient is fluent in English
* patient taking newly-prescribed antidepressant for no more than 1 week

Exclusion Criteria:

* patient with plans of leaving the vicinity within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2006-07; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Persistence

SECONDARY OUTCOMES:
Adherence (mean possession ratio)
Beck Depression Inventory symptom improvement
Beck Anxiety Inventory symptom improvement
Change in antidepressant compliance questionnaire responses

CONTACTS AND LOCATIONS:
Overall Officials: David M Gardner, PharmD, Principal Investigator — Dalhousie University
Locations (1):
- EPICORE Centre, Edmonton, Alberta, Canada